CLINICAL TRIAL: NCT02613559
Title: A Single-center, Open-label, Single Ascending Dose Phase 1 Study to Evaluate the Safety, Pharmacokinetics, and Tolerability of Intravitreal TK001(Recombinant Humanized Anti-VEGF Monoclonal Antibody) in Subjects With Neovascular Age-Related Macular Degeneration
Brief Title: Evaluation the Pharmacokinetics, Safety, Tolerability of TK001 in Patients With Neovascular Age-related Macular Degeneration
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu T-Mab Biopharma Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tmab-TK001-AMD-01
Record Dates: First submitted 2015-11-21; First posted 2015-11-24 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Neovascular Age-Related Macular Degeneration, Subfoveal CNV, TK001

ARMS (6):
- TK001 0.1mg (Experimental): Injection:single Intravitreal Injection
  Interventions: Biological: TK001
- TK001 0.5mg (Experimental): Injection:single Intravitreal Injection
  Interventions: Biological: TK001
- TK001 1.0mg (Experimental): Injection:single Intravitreal Injection
  Interventions: Biological: TK001
- TK001 2.0mg (Experimental): Biological: TK001 Injection:single Intravitreal Injection
  Interventions: Biological: TK001
- TK001 2.5mg (Experimental): Biological: TK001 Injection:single Intravitreal Injection
  Interventions: Biological: TK001
- TK001 3.0mg (Experimental): Injection:single Intravitreal Injection
  Interventions: Biological: TK001

INTERVENTIONS:
Biological: TK001 — Intravitreal Injection

SUMMARY:
The purpose of this first-in-human study is to evaluate the safety, pharmacokinetics and tolerability of single ascending doses of TK001(Recombinant humanized anti-VEGF monoclonal antibody) to determine the maximum tolerated dose (MTD) in neovascular wet age-related macular degeneration (wAMD) subjects.

DETAILED DESCRIPTION:
This is an open-label, non-comparative, non-randomized, single-center phase 1 study evaluating pharmacokinetics, safety and tolerability of single intravitreal injections of TK001 in the patients with AMD.TK001 is a full-length recombinant humanized anti-VEGF monoclonal antibody. Compared with Avastin(a similar marketed product), the findings of preclinical studies suggested that TK001 might be more effective in inhibiting pathological angiogenesis, or to achieve equivalent effect with less dosage and better safety. In this study, participants will be administrated a single dose of TK001.Every subject will only accept one dose. In addition to safety and preliminary efficacy, pharmacokinetics and immunogenicity of TK001will be evaluated as well.

ELIGIBILITY:
Inclusion Criteria:

* Patients or their legal representative signed informed consent
* Aged 45 years to 80 years, male or female
* Inpatient/Outpatient with confirmed neovascular AMD
* Best corrected VA for the studied eye≤20/100
* With primary or recurrent subfoveal choroidal neovascular (CNV) lesions secondary to neovascular AMD
* Blood pressure is stable with SBP<140 mmHg and DBP<90 mmHg with or without treatment

Exclusion Criteria:

* Limitation of eye diseases

  1. The studied eye suffered intravitreal blood within two months prior to screening
  2. The studied eye suffered structural damage of retinal which involved macular center(such as epiretinal membrane, scars, laser burns, foveal atrophy, dense pigment changes, intensive subfoveal hard exudates)
  3. Apparent cataract, aphakia, pseudoexfoliation syndrome, intraocular hemorrhage resulting in decreased vision, rhegmatogenous retinal detachment, macular hole, diabetic retinopathy and diabetic macular disease which need to be treated, choroidal neovascularization (CNV) for any reason except for AMD (such as ocular histoplasmosis, pathologic myopia)
  4. Afferent pupillary defect(APD)
  5. Refractive media opacity and miosis which effect fundus examination
  6. Any eye of patient with active inflammation, such as conjunctivitis, keratitis, scleritis, uveitis and endophthalmitis
  7. Choroidal neovascularization (CNV) for other reason, such as diabetic retinopathy, fundus angioid streaks, ocular histoplasmosis, pathologic myopia, trauma
* The treatment of the eye

  1. The studied eye received topical or grid photocoagulation more than twice or within 3 months before screening
  2. The studied eye received any intraocular surgery or laser treatment (such as macular translocation surgery, glaucoma filtering surgery, verteporfin photodynamic therapy, transpupillary thermotherapy, foveal photocoagulation surgery, cataract surgery, vitreous cutting surgery, optic nerve incision operation, YAG posterior capsular incision surgery, sheath incision surgery or filtering surgery) within 3 months before screening
  3. Any eye received antiangiogenic drugs (including any anti-VEGF drugs) (such as pegaptanib [Macugen®], Aflibercept [Eylea®], ranibizumab [Lucentis ®], bevacizumab [Avastin ®]) within 3 months before baseline visit
  4. Any eye received intraocular injection of corticosteroid drugs (such as triamcinolone acetonide), or periocular injection of corticosteroid drugs within 1 months before screening
* Systemic diseases,treatment and other conditions

  1. With a history of allergy to sodium fluorescein and indocyanine green
  2. PLT≤100×109/L, BUN, Cr, thrombin time and prothrombin time beyond the upper limit of the normal range; take anti-platelet aggregation drugs within a month prior to enrollment
  3. With surgery within one month prior to enrollment, or with unhealing wound, ulcer, fracture at present
  4. Diabetic patients without the control of glucose or accompanied by diabetic retinopathy
  5. With a history of myocardial infarction within 6 months before enrolled
  6. With activity disseminated intravascular coagulation and a tendency of significant bleeding prior to enrollment
  7. Systemic autoimmune disease
  8. Any uncontrolled clinical problems (such as severe systemic diseases of mental, neurological, cardiovascular, respiratory and malignancies)
  9. Pregnant and lactating women and patients who cannot take contraceptive measures
  10. Poor compliance
  11. The patients who is considered unsuitable for enrollment by investigator

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-06 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Frequency of ocular and systemic AEs (adverse events) and SAEs (serious adverse events) which are related to TK001 | 6 weeks

SECONDARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) | 6 weeks
Area under the plasma concentration-time curve from time zero to infinity (AUCinf) | Up to Day 42
Area under the plasma concentration-time curve from time zero to time 't' where t is a defined time point after administration (AUC0-t) | Up to Day 42
Maximum observed maximum plasma concentration (Cmax) | Up to Day 42
Time to reach the maximum observed plasma concentration (Tmax) | Up to Day 42
Frequency of subjects with anti-TK001 antibody | Up to Day 42
  Anti- TK001 antibody will be detected pre-dose,14d and 42d.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhang, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China